CLINICAL TRIAL: NCT07035860
Title: Efficacy and Safety of Induction Chemoimmunotherapy Followed by Carbon Ion Radiotherapy and Consolidation Immunotherapy in Unresectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Chemoimmunotherapy and Carbon Ion Radiotherapy in Unresectable Locally Advanced Non-small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Ji Yongling (Other)
Responsible Party: Sponsor-Investigator, Ji Yongling, PI, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: HZCIRT-Lung 001
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Carbon Ion Radiotheray
Keywords: non-small cell lung cancer; carbon ion radiotherapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Heavy Ion Radiotherapy; Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue, blood, urine, and stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Induction chemoimmunotherapy followed by carbon ion radiotherapy and consolidation immunotherapy
  Interventions: Radiation: Carbon ion radiotherapy; Drug: Chemotherapy; Drug: Immunotherapy

INTERVENTIONS:
Radiation: Carbon ion radiotherapy — Patients will receive platinum-based doublet chemotherapy and immunotherapy, followed by carbon iron radiotherapy and immunotherapy. The concrete immune checkpoint inhibitor includes durvalumab, sugemalimab, atezolizumab, benmelstobart, pembrolizumab, camrelizumab, toripalimab, tislelizumab, sintilimab, nivolumab, serplulimab, or penpulimab.
Drug: Chemotherapy — platinum-based doublet chemotherapy
Drug: Immunotherapy — The concrete immune checkpoint inhibitor includes durvalumab, sugemalimab, atezolizumab, benmelstobart, pembrolizumab, camrelizumab, toripalimab, tislelizumab, sintilimab, nivolumab, serplulimab, or penpulimab.

SUMMARY:
This is the first prospective clinical study to evaluate the efficacy and safety of induction chemoimmunotherapy followed by carbon ion radiotherapy and consolidation immunotherapy in patients with unresectable locally advanced non-small cell lung cancer (NSCLC). Based on this prospective study, tumor tissue, blood, urine, and stool samples from participants will be collected and analyzed to identify predictive markers of treatment response.

DETAILED DESCRIPTION:
All patients had a pathologically confirmed locally advanced NSCLC according to the 8th AJCC staging system would receive platinum-based doublet chemotherapy and immunotherapy, followed by carbon iron radiotherapy and immunotherapy. The concrete immune checkpoint inhibitor includes durvalumab, sugemalimab, atezolizumab, benmelstobart, pembrolizumab, camrelizumab, toripalimab, tislelizumab, sintilimab, nivolumab, serplulimab, or penpulimab.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced non-small cell lung cancer (according to the 8th edition of the AJCC staging system).
* No prior anti-cancer treatment.
* No significant internal medical conditions or major organ dysfunction.

Exclusion Criteria:

* Histological evidence of small cell lung cancer or other primary malignancies
* EGFR, ALK, or ROS-1 gene mutations.
* Active or prior autoimmune/inflammatory disorders.
* Inability to comply with study protocol as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable locally advanced non-small cell lung cancer (according to the 8th edition of the AJCC staging system).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
1-year PFS | 12 months
  Time between enrollment and recurrence of disease or death
Incidence of Grade ≥3 Treatment-Related Adverse Events | Occurrence or end of follow-up（3 years after enrollment), which comes first
  Safety

SECONDARY OUTCOMES:
OS | Occurrence or end of follow-up（3 years after enrollment）, which comes first
  Time between enrollment and death

OTHER OUTCOMES:
Biomarker Analysis | 36 months
  Including ctDNA levels and their correlation with treatment response; additional biomarkers include PD-L1 expression, TMB, RNA expression profiles, immune cell subtypes, cytokines, metabolites, tumor and gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Yongling JI, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No